CLINICAL TRIAL: NCT03064919
Title: Developing Novel Methods to Teach Children to Recognize Internal Signals of Hunger and Fullness
Brief Title: Developing Novel Methods to Teach Children to Recognize Internal Signals of Hunger
Acronym: CTSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Director, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Hunger and Fullness
Record Dates: First submitted 2017-02-01; First posted 2017-02-27 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Obesity
Keywords: hunger and fullness; regulation of energy intake; energy compensation; nutrition knowledge
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: An evidence-based curriculum for teaching preschool children to eat in response to internal hunger and fullness signals will be developed. The investigators will then conduct an experimental study to determine the effectiveness of this curriculum on children's ability to regulate energy intake in the laboratory. Key outcomes will be children's adjustment in intake in response to a first course (energy compensation) and children's intake of tasty snacks when not hungry (eating in the absence of hunger). Data describing variables likely to impact the success of the curriculum will be collected, for example: child gender/age, parent feeding practices, parent education, infant feeding practices, child/parent weight status, and others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curriculum Testing (Experimental): Test an evidence-based curriculum for teaching preschool children to eat in response to internal hunger and fullness signals.
  Interventions: Behavioral: Curriculum Testing

INTERVENTIONS:
Behavioral: Curriculum Testing — An evidence-based curriculum for teaching preschool children to eat in response to internal hunger and fullness signals was developed by refining an existing curriculum. State-of-the art theories in early childhood science education, innovative virtual technology to provide more realistic simulations of hunger and fullness, and a parent training component to improve long-range sustainability were incorporated. This 9-wk intervention will be tested by forty children (ages 4-5). Key outcomes will be children's adjustment in intake in response to a first course (energy compensation) and children's intake of tasty snacks when not hungry (eating in the absence of hunger). Additionally, the investigators will measure other variables likely to impact the success of the curriculum, for example: child gender/age, parent feeding practices, parent education, infant feeding practices, child/parent weight status, and others.

SUMMARY:
The purpose of this multi-year project is to develop an evidence-based curriculum for teaching preschool children to eat in response to internal hunger and fullness signals. There are currently no validated methods for teaching children these basic skills, despite the fact that doing so is necessary to prevent the development of obesity.

DETAILED DESCRIPTION:
The purpose of this multi-year project is to develop an evidence-based curriculum for teaching preschool children to eat in response to internal hunger and fullness signals. There are currently no validated methods for teaching children these basic skills, despite the fact that doing so is necessary to prevent the development of obesity. To accomplish this task, the investigators have assembled a multi-disciplinary team from nutrition, eating behavior, obesity prevention, science education, and information sciences and technology.

First, the investigators will refine and build upon a pre-existing curriculum by incorporating 1) state-of-the art theories in early childhood science education, 2) innovative virtual technology to provide more realistic simulations of hunger and fullness, and 3) a parent training component to improve long-range sustainability.

Second, the investigators will conduct an experimental study to determine the effectiveness of this curriculum on children's ability to regulate energy intake in the laboratory. Forty children (ages 4-5) will be tested over an 9-week period. Key outcomes will be children's adjustment in intake in response to a first course (energy compensation) and children's intake of tasty snacks when not hungry (eating in the absence of hunger). Additionally, the investigators will measure other variables likely to impact the success of the curriculum, for example: child gender/age, parent feeding practices, parent education, infant feeding practices, child/parent weight status, and others.

The long term goal of this line of research will be to create an evidence based curriculum that can be integrated into early childhood education and health-based interventions. The translation potential of this research is broad because once validated, the curriculum can be disseminated more widely to early childhood education programs.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between the ages of 4-5 years-old at the time they participate in the study.
* All children will be physically healthy, with no food allergies. Parents are asked if the child has any medical problems or is taking any prescription medication. If the answer to either of these questions is yes but the medical problem (or medication) is not severe nor has the potential to affect the study outcome, as judged by our PI, then the child may be included.
* The person primarily responsible for feeding the child must be able to make nine, two-hour visits along with the child to the lab within an nine-week time period.

Exclusion Criteria:

* Child is younger than 4 or older than 6.
* Child is not physically healthy. Parents are asked if the child has any medical problems or is taking any prescription medication. If the medical problem (or medication) is severe or may affect the study outcome, as judged by our PI, then the child may be excluded.
* Child has food allergies.
* Person primarily responsible for feeding child and child cannot make nine, 90 minute - 2 hour visits along with the child within a 9-week period.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Energy Compensation measured by compensation score. | Change from baseline to 9 weeks later.
  Children's ability to compensate for calories in a first course will be assessed by measurement of compensation score. The Compensation Score will be measured over two baseline lab sessions where children are served a low-energy drink (~3 calories) or a high-energy drink (150 calories), followed 25-30 minutes later by a buffet test-meal consisting of the common foods listed above.
Eating in the Absence of Hunger after a buffet meal: Food Intake weighed in grams and calories. | Change from baseline to 9 weeks later.
  Children's intake (grams and calories) of tasty snacks when not hungry (eating in the absence of hunger). This measurement is taken after a buffet meal is served.
Energy intake at a buffet meal | Change from baseline to 9 weeks later
  Measured at an objective laboratory test meal (kcal and grams)
Nutrition knowledge test for children | Change from baseline to 9 weeks later
  Age appropriate nutrition questions, with questions such as: 1) What body parts are involved with digestion? 2) Why do we eat? 3) Why do we stop eating? 4) What happens when we eat too much? and 5) Simulation of eating just the right amount using a computer game.

SECONDARY OUTCOMES:
Liking of foods | Baseline and 9 weeks later.
  Ratings of how much a child likes specific foods used in the study test meals, completed on visual analog scales.
Wanting of foods | Baseline and 9 weeks later.
  Ratings of how much a child wants to eat specific foods used in the study test meals, completed on visual analog scales.
Fullness feelings | Baseline and 9 weeks later.
  Ratings of how full the child feels on a child friendly visual analog scale.
Height | Baseline and 9 weeks later.
  Height in m measured by a stadiometer.
Weight | Baseline and 9 weeks later.
  Weight in kg by standard digital scale.
Body mass index | Baseline and 9 weeks later.
  Calculated from height and weight (kg/m^2)
BMI percentile | Baseline and 9 weeks later.
  Calculated from height, weight, age, sex
BMI z-score | Baseline and 9 weeks later.
  Calculated from height, weight, age, sex
Child Eating Behavior Questionnaire | Baseline and 9 weeks later.
  Parent-reported questionnaire of habitual eating styles in children.
Pubertal development Questionnaire | Baseline
  Parent-reported questionnaire
Family demographics | Baseline
  Parent-reported questionnaire
Child feeding Questionnaire | Baseline and 9 weeks later.
  Parent-reported questionnaire of feeding strategies.
Infant Feeding Questionnaire | Baseline and 9 weeks later.
  Parent-reported questionnaire of infant feeding.
Child Behavior | Baseline and 9 weeks later.
  Parent-reported questionnaire of child behavior.
Parent Eating Competence | Baseline and 9 weeks later.
  Parent-reported questionnaire of parent eating competence.
Division of Responsibility in Child Feeding Questionnaire | Baseline and 9 weeks later.
  Parent-reported questionnaire of division of responsibility in child feeding
Nutrition Steps Questionnaire | Baseline and 9 weeks later.
  Standardized nutrition questionnaire.
Caregiver Feeding Style Questionnaire | Baseline and 9 weeks later.
  Parent-reported questionnaire of caregiver feeding style

OTHER OUTCOMES:
Child Age | Baseline
  Child age in months.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No